CLINICAL TRIAL: NCT05808296
Title: The Effect of Lavender Oil on Fatigue and Sleep Quality in Patients With Hematologic Malignancy: A Single Blinding Randomized Controlled Study
Brief Title: The Effect of Lavender Oil on Fatigue and Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Prof., Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Lavender Oil on Hematological
Record Dates: First submitted 2023-03-30; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Hematologic Malignancies; Patient Participation
Keywords: Sleep Disorders; Aroma Therapy; Hematologic Malignancies; Fatigue
MeSH Terms: conditions — Hematologic Neoplasms; Patient Participation; Sleep Wake Disorders; Fatigue | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): aromatherapy will be performed by dropping 2 drops of lavender oil on the shoulder with a sponge 20 minutes before bedtime every night for a week
  Interventions: Other: Lavander oil Aromatherapy
- Control (Sham Comparator): Saline solution will be performed by dropping 2 drops of saline solution on the shoulder with a sponge 20 minutes before bedtime every night for a week
  Interventions: Other: Saline Solution

INTERVENTIONS:
Other: Lavander oil Aromatherapy — Lavander oil Aromatherapy
  Arms: Experiment
Other: Saline Solution — Saline solution application
  Arms: Control

SUMMARY:
This study will be conducted in a randomized, controlled and experimental manner with patients with hematological malignancies admitted to the Adult Bone Marrow Transplant unit and Hematology-Oncology unit of Acıbadem Altunizade Hospital after obtaining the necessary permissions. The number of patients to be included in the study will be determined by power analysis. The study will include patients who are willing to participate, have no communication problems, are 18 years of age or older, and have no known allergy to lavender oil. Patients with allergies, drug addiction and refusal to participate in the study will not be included in the study. Before the study, patients will be divided into intervention and control groups using a simple random number table. At the beginning of the study, a form including socio-demographic and disease information, Richard Campbell Sleep Quality Scale and Piper Fatigue Scale will be evaluated. Two different options will be used to prevent findings. The first group will be treated with lavender oil and the second group will be treated with saline and 2 drops will be placed on the patient's shoulder 20 minutes before bedtime every night. The application will be started simultaneously with the chemotherapy and will continue until the end of chemotherapy treatment. Sleep and fatigue will be assessed daily using the Richard Campbell Sleep Quality Scale and Piper Fatigue Scale.

DETAILED DESCRIPTION:
Insomnia and fatigue symptoms, which are common in patients with hematologic malignancies, affect the quality of life of patients and may increase the severity of other symptoms. Pharmacologic and non-pharmacologic methods can be used in the management of insomnia and fatigue. Nonpharmacologic approaches are also used because pharmacologic methods have side effects and their effects on sleep and fatigue are not fully proven. One of the nonpharmacological approaches used is lavender oil inhalation. The effects of lavender oil on sleep and fatigue have been shown in studies. In addition, no national or international study results evaluating the effect of lavender oil on fatigue and sleep quality in patients with hematologic malignancy were found in the literature. Based on this, the study was planned to examine the effect of lavender oil on sleep quality and vital signs of palliative care patients.

This study will be conducted in a randomized, controlled and experimental manner with patients with hematological malignancies admitted to the Adult Bone Marrow Transplant unit and Hematology-Oncology unit of Acıbadem Altunizade Hospital after obtaining the necessary permissions. The number of patients to be included in the study will be determined by power analysis. The study will include patients who are willing to participate, have no communication problems, are 18 years of age or older, and have no known allergy to lavender oil. Patients with allergies, drug addiction and refusal to participate in the study will not be included in the study. Before the study, patients will be divided into intervention and control groups using a simple random number table. At the beginning of the study, a form including socio-demographic and disease information, Richard Campbell Sleep Quality Scale and Piper Fatigue Scale will be evaluated. Two different options will be used to prevent findings. The first group will be treated with lavender oil and the second group will be treated with saline and 2 drops will be placed on the patient's shoulder 20 minutes before bedtime every night. The application will be started simultaneously with the chemotherapy and will continue until the end of chemotherapy treatment. Sleep and fatigue will be assessed daily using the Richard Campbell Sleep Quality Scale and Piper Fatigue Scale.

Statistical Package for Social Science (SPSS) statistical package program will be used in the evaluation of the data, the conformity of the data to normal distribution will be questioned with Kollmogorov Smirnov test, mean, standard deviation, correlation values will be examined and T-Test will be used to evaluate the relationship between independent groups.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study and being 18 years of age or older
* Cooperation, no communication problems
* Systolic blood pressure above 100 mmHg (lavender can cause hypotension)
* Staying in the bone marrow transplant service for at least two days

Exclusion Criteria:

* Known diagnosis of a psychiatric illness (anxiety, panic attacks, depression), a known history of allergy and use of anxiolytic drugs.
* Having arrhythmia
* Do not use sleeping pills
* Allergy to any essential oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive information form | 1. day.
  The form includes demographic data such as age, gender and education level
Richards Campbell Sleep Quality Scale (RCSQ) | 1. day
  The sleep quality of the patients was evaluated three times with the Richards Campbell Sleep Quality Scale: preintervention, postintervention day 1 and postintervention day 2. The Richards Campbell Sleep Quality Scale consists of six items evaluating the depth of the patients' night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep and the noise level in the environment. Each item is evaluated by the patient by questioning the patient's night sleep on a visual analog scale of 0-100. The total score of the scale is obtained from the sum of the five items. The 6th item evaluating the ambient noise level is excluded from the total score evaluation. A score between "0-25" indicates that the quality of the patient's night sleep is very poor and a score between "76-100" indicates that the quality of the patient's night sleep is very good.
Richards Campbell Sleep Quality Scale (RCSQ) | 7. day
  The sleep quality of the patients was evaluated three times with the Richards Campbell Sleep Quality Scale: preintervention, postintervention day 1 and postintervention day 2. The Richards Campbell Sleep Quality Scale consists of six items evaluating the depth of the patients' night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep and the noise level in the environment. Each item is evaluated by the patient by questioning the patient's night sleep on a visual analog scale of 0-100. The total score of the scale is obtained from the sum of the five items. The 6th item evaluating the ambient noise level is excluded from the total score evaluation. A score between "0-25" indicates that the quality of the patient's night sleep is very poor and a score between "76-100" indicates that the quality of the patient's night sleep is very good.
Piper Fatigue Scale | 1. day
  The scale developed by Piper B. F. et al. in 1998 consists of a total of 22 items and evaluates the patient's subjective perception of fatigue with four sub-dimensions. These are the behavior/severity sub-dimension (6 items; 2-7), which evaluates the impact and severity of fatigue on activities of daily living (ADL); the affect sub-dimension (5 items; 8-12), which covers the emotional meaning attributed to fatigue; the sensory sub-dimension (5 items; 13-17), which reflects the mental, physical and emotional symptoms of fatigue; and the cognitive/mental sub-dimension (6 items; 18-23), which reflects the level of fatigue affecting cognitive functions and mental state. In addition, there are 5 items (1 and 24-27).
Piper Fatigue Scale | 7. day
  The scale developed by Piper B. F. et al. in 1998 consists of a total of 22 items and evaluates the patient's subjective perception of fatigue with four sub-dimensions. These are the behavior/severity sub-dimension (6 items; 2-7), which evaluates the impact and severity of fatigue on activities of daily living (ADL); the affect sub-dimension (5 items; 8-12), which covers the emotional meaning attributed to fatigue; the sensory sub-dimension (5 items; 13-17), which reflects the mental, physical and emotional symptoms of fatigue; and the cognitive/mental sub-dimension (6 items; 18-23), which reflects the level of fatigue affecting cognitive functions and mental state. In addition, there are 5 items (1 and 24-27).

CONTACTS AND LOCATIONS:
Locations (1):
- Dilek Yildirim, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yildirim D, Harman Ozdogan M, Erdal S, Selcuk S, Guneri A, Simsek EB, Can TB, Gunduz H, Kuni A. The efficacy of lavender oil on fatigue and sleep quality in patients with hematological malignancy receiving chemotherapy: a single-blind randomized controlled trial. Support Care Cancer. 2025 Jan 8;33(2):79. doi: 10.1007/s00520-024-09143-5. PMID 39775962